CLINICAL TRIAL: NCT00161226
Title: A Randomized, Controlled, Comparative Study of a Levonorgestrel Intrauterine System for the Prevention of Endometrial Cancer in Patients Aged 40-50 With BMI Greater Than 35
Status: Terminated | Type: Observational
Why Stopped: Principal investigator left institution
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 4800; CINJ#100401
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: Levonorgestrel intrauterine system

SUMMARY:
Endometrial (uterine) cancer affects over 40,000 women each year in the United States. At this time there are no medications to prevent endometrial cancer. Women who are heavy are at increased risk of this cancer. Progestins have been used to treat endometrial hyperplasia and cancer in women who wanted to retain their fertility or who were not surgical candidates. Oral progestins are associated with side effects such as weight gain, mood changes, headaches, and acne. A device called Mirena has a type of progesterone in it. Because it is placed directly in the uterus it can give a powerful amount of progestin with less side effects. In this project, we will enroll 44 women who are aged 40-50 and who have a body mass index (BMI) greater than 40. (BMI is a measure of obesity. Normal is less than 25.) They will be randomized to either observation or treatment. The women in the treatment group will have a levonorgestrel intrauterine system (Mirena, LNG-IUS) placed for one year. All of the women will have endometrial biopsies and blood work at the beginning and end of the study. All of the women will have an ultrasound at the beginning of the study. The information will then be used to assess whether or not the LNG-IUS will be an effective prevention agent. The women will be contacted once a year for 5 years to see if they have had endometrial hyperplasia or cancer. A special lab study called microarray will be used to see what genes are turned on or off in the uterine lining.

DETAILED DESCRIPTION:
Endometrial (uterine) cancer affects over 40,000 women each year in the United States. At this time there are no medications to prevent endometrial cancer. Women who are heavy are at increased risk of this cancer. Progestins have been used to treat endometrial hyperplasia and cancer in women who wanted to retain their fertility or who were not surgical candidates. Oral progestins are associated with side effects such as weight gain, mood changes, headaches, and acne. A device called Mirena has a type of progesterone in it. Because it is placed directly in the uterus it can give a powerful amount of progestin with less side effects. In this project, we will enroll 44 women who are aged 40-50 and who have a body mass index (BMI) greater than 40. (BMI is a measure of obesity. Normal is less than 25.) They will be randomized to either observation or treatment. The women in the treatment group will have a levonorgestrel intrauterine system (Mirena, LNG-IUS) placed for one year. All of the women will have endometrial biopsies and blood work at the beginning and end of the study. All of the women will have an ultrasound at the beginning of the study. The information will then be used to assess whether or not the LNG-IUS will be an effective prevention agent. The women will be contacted once a year for 5 years to see if they have had endometrial hyperplasia or cancer. A special lab study called microarray will be used to see what genes are turned on or off in the uterine lining.

ELIGIBILITY:
Inclusion:

Woman between 40-50 years of age. Body mass index (BMI) ³ 35. Benign (no hyperplasia or cancer) endometrial biopsy prior to randomization Has an intact uterus

Exclusion:

Present infection with gonorrhea or chlamydia or within the last 5 years. Bacterial vaginosis that does not respond to one course of antibiotics. History of pelvic inflammatory disease in the last 5 years. Patients who are pregnant or who desire to become pregnant Does not desire fertility History of deep venous thrombosis or pulmonary embolus

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Levonorgestrel IUD, Prevention of Endometrial Cancer, Patients Aged 35-50, BMI > 30
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2004-02; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Wagreich, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States